CLINICAL TRIAL: NCT00557765
Title: Production of Gamma-Interferon by Circulating Lymphocytes Exposed to Antigens Specific of Mycobacterium Tuberculosis: Contribution to the Identification of Latent Tuberculosis Infection in Contact Tracing
Brief Title: Use of a Gamma-IFN Assay in Contact Tracing for Tuberculosis in a Low-Incidence, High Immigration Area
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: Ligue Pulmonaire Genevoise (Other)
Other Study IDs: 04-184
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-11

CONDITIONS: Tuberculosis; Latent Tuberculosis Infection
Keywords: Tuberculosis; Latent tuberculosis infection; Interferon gamma release assay; Contact tracing
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
After exposure to an active case of tuberculosis (TB), close contacts may be infected. They are then considered as having latent tuberculosis infection (LTBI). Detecting LTBI is the main goal of contact tracing procedures after exposure to TB. Until recently, the only test available for detecting LTBI was the tuberculin skin test (TST). More recent tests are now available (Interferon-gamma release assays: IGRA), which are more specific and sensitive than the TST. This study compares the TST and an IGRA in the routine activity of contact tracing in our area.

DETAILED DESCRIPTION:
Setting: A TB clinic in Geneva, Switzerland, a low incidence area for TB with a high immigrant population.

Aim of study: to compare results of an IGRA test (T-SPOT.TB, Oxford Immunotec, UK) and the TST, and their correlation with exposure scores in subjects exposed to cases of contagious TB.

Methods: Prospective study of all contacts screened in our area, and accepting to be included. Simultaneous recording of age, gender, origin, history of recent travels or exposure, BCG vaccination status, infectiousness of index case, 5 different exposure scores, TST, and result of the T-SPOT.TB blood test. Univariate and multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* Exposure to a case of contagious TB
* Willingness to participate in study

Exclusion Criteria:

* Known HIV infection
* Known previous TB or treatment for LTBI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects screened after exposure to a case of active and contagious tuberculosis in the Geneva area
Sampling Method: Non-Probability Sample
Enrollment: 295 (Actual)
Dates: Start 2004-10; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Correlation between results of TST and IGRA tests and exposure scores | 2 months after exposure

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Janssens, M.D., Principal Investigator — Centre antituberculeux
Locations (1):
- Centre antituberculeux; Geneva University Hospital, Geneva, Canton of Geneva, Switzerland